CLINICAL TRIAL: NCT02033967
Title: Vasodilator-induced Hypovolemia in Living Liver Donors: Central Venous Pressure-guided vs Stroke Volume Variation-guided Technique
Brief Title: Vasodilator-induced Hypovolemia in Living Liver Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chul-Woo Jung, associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MLN_SVV_CVP
Record Dates: First submitted 2014-01-08; First posted 2014-01-13 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: CVP and SVV During Living Donor Hepatectomy; Surgical Field Grade (Condition of Surgical Field; Bleeding, Tension of the IVC)
Keywords: liver donor; hepatectomy; vasodilator; central venous pressure; stroke volume variation
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CVP (Active Comparator): Central venous pressure-guided vasodilator-induced hypovolemia
  Interventions: Procedure: vasodilator induced hypovolemia
- SVV (Experimental): stroke volume variation-guided vasodilator-induced hypovolemia
  Interventions: Procedure: vasodilator induced hypovolemia

INTERVENTIONS:
Procedure: vasodilator induced hypovolemia
  Other Names: Milrinone induced hypovolemia

SUMMARY:
Induced hypovolemia is known to improve surgical field during living donor hepatectomy. This procedure is conventionally guided by monitoring the central venous pressure (CVP). Stroke volume variation (SVV) is a novel method to substitute with CVP to monitor cardiac preload. The investigators try to evaluate the relationship between CVP and SVV during CVP-guided vasodilator induced hypovolemia (validation study). Then, feasibility of vasodilator induced hypovolemia using the SVV calculated from the validation study will be tested (feasibility study).

DETAILED DESCRIPTION:
This is a 2-phases study.

first phase validation study : Evaluation of the relationship between CVP and SVV during CVP-guided vasodilator induced hypovolemia

second phase feasibility study

: Comparison of the surgical field grade between validation study group(CVP guided group) and feasibility study group(SVV guided group)

ELIGIBILITY:
Inclusion Criteria:

* adult (20-60 yr)
* elective living liver donors

Exclusion Criteria:

* not obtained informed consent

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
target value of SVV | during living donor hepatectomy
  Target value of SVV is calculated from the linear regression equation that was calculated from scatter plot made with CVP and SVV values during CVP-guided vasodilator induced hypovolemia (validation study).

SECONDARY OUTCOMES:
surgical field | during living donor hepatectomy
  <4 point scale> Grade l: Very lax IVC and hepatic veins, minimal bleeding at resection plane, very easy to operate Grade ll: Lax IVC and hepatic veins, a little bleeding at resection plane, easy to operate Grade lll: Tense IVC and hepatic veins, appreciable bleeding at resection plane, somewhat difficult to operate Grade lV: Very tense IVC and hepatic veins, profuse bleeding at resection plane, very difficult to operate
use of inotropics | during living donor hepatectomy
estimated blood loss | during living donor hepatectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee J, Kim WH, Ryu HG, Lee HC, Chung EJ, Yang SM, Jung CW. Stroke Volume Variation-Guided Versus Central Venous Pressure-Guided Low Central Venous Pressure With Milrinone During Living Donor Hepatectomy: A Randomized Double-Blinded Clinical Trial. Anesth Analg. 2017 Aug;125(2):423-430. doi: 10.1213/ANE.0000000000002197. PMID 28632543